CLINICAL TRIAL: NCT01144650
Title: Clinical Trial Randomized, Placebo-controlled, Using Dapsone as a Neuroprotector During Acute Ischemia Stroke
Brief Title: Dapsone for Acute Ischemia Stroke Study
Acronym: DAISY
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cidat, S.A. de C.V. (Industry)
Collaborators: El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez (Other)
Responsible Party: Camilo Rios, PhD, Instituto Nacional de Neurologia y Neurocirugia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIDAT-072009-DAA-MC
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-06

CONDITIONS: Cerebral Stroke; Cerebrovascular Accident, Acute; Cerebrovascular Stroke; Stroke, Acute; Stroke
Keywords: Dapsone; Cerebrovascular Accident, Acute; Neuroprotection
MeSH Terms: conditions — Stroke | interventions — Dapsone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients will receive either a single total dose of 250 mg placebo IV and oral dosage
  Interventions: Drug: Placebo
- Dapsone (Experimental): Patients will receive either a single total dose of 250 mg IV and oral dosage
  Interventions: Drug: Dapsone

INTERVENTIONS:
Drug: Dapsone — Patients will receive either a single total dose of 250 mg dapsone or placebo IV and oral dosage
  Other Names: diamino-diphenyl sulfone; DDS
  Arms: Dapsone
Drug: Placebo — Patients will receive either a single total dose of 250 mg placebo IV and oral dosage
  Arms: Placebo

SUMMARY:
The main purpose of the study is to get information about the safety and efficacy of treatment with Dapsone to prevent the disability after ischemic Stroke, in patients diagnosed with anterior territory brain infarct.

DETAILED DESCRIPTION:
Cerebrovascular diseases are the third cause of mortality around the world. Seventy-five percent of the cases correspond to ischemic stroke, and the remaining 25 % to hemorrhagic infarct. The social impact of Stroke is high as it is the first cause for disabilities. After Stroke, several mechanisms of secondary damage act to spread the damage to the surrounding tissue. Those mechanisms include: 1) Excitotoxicity after excitatory amino acids' release 2) Overproduction of free radicals 3) Exacerbated inflammatory response and 4) Apoptosis. Many neuroprotective strategies have been tested to cope with the already mentioned damaging processes with poor clinical results. Many clinical trials have failed to provide neuroprotection to patients after acute stroke. Then, the need for safe drugs with clinical efficacy to prevent Stroke disability consequences is highly recognized. Dapsone is safe and relatively free of adverse reactions, we propose a clinical trial to assess the safety and efficacy of using this drug in patients with ischemic brain stroke.

Methods: A double-blind, placebo-controlled, randomized clinical trial of dapsone is to be conducted from 2009 to 2010. Three-hundred patients with a CT or MRI documented ischemic stroke in the anterior cerebral territory are to be included. Patients with 4 to 20 points of the National Institute of Health Stroke Scale (NIHSS) will be randomly allocated to receive either a single total dose of 250 mg dapsone or placebo within the first 12 h after stroke. For the follow-up, NIHSS on days 0, 2, 7, 30, 60 and 90, modified Rankin scale (mRS) on days 0, 30, 60 and 90, and Barthel index (BI) at day 90, will be all applied. Adverse reactions will be also recorded. The Primary clinical outcome of the patients will be assessed at 90 days after stroke by obtaining the shift analysis from the baseline levels of the scales mRS and NIHSS. Secondary clinical outcome will be the BI at day 90. An interim analysis of the data will be performed when the study have recruited one-hundred patients.

Statistical analysis will be performed with the intention-to-treat approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the clinical diagnosis of an acute cerebrovascular event in in the anterior cerebral territory, within the last 12 hours who match the MRI or axial CT image.
* Patients with 4 o more points of the National Institute of Health Stroke Scale (NIHSS)
* Age older than 18 years, both gender
* Non acute cerebrovascular event previous
* Informed consent signed by patient or relatives

Exclusion Criteria:

* Diagnosed with recurrent diseases like: heart failure; Myocardial Infarction up 8 weeks before; ventrivular arrhythmia diagnosed by ECG; Second-Degree and Third-Degree Atrioventricular Block; or Long QT Syndrome.
* Pregnancy
* Allergic reactions to sulfa medications
* Patients with kidney failure and hepatic insufficiency
* Deficiency of glucose-6-phosphate dehydrogenase diagnosed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-08 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Shift across the board of National Institute of Health stroke scale (NIHSS) and Modified Rankin Scale (mRS) | 90 days after stroke
  The NIHSS is a deficit severity scale that assigns 42 points to patients according to the degree of neurologic deficits.
  The mRS is a severity scale for the assessment of global disability into 7 points: 0= no disability,1=non-significant disability, 2=slight disability, 3=moderate disability, 4= moderately severe disability, 5= severe disability, 6= dead

SECONDARY OUTCOMES:
Barthel index | 90 days after stroke
  The Barthel Index evaluates the daily-live activities rating in 20 points of functional activities.

CONTACTS AND LOCATIONS:
Overall Officials: Juan A. Nader, MD, Principal Investigator — Hospital Medica Sur
Locations (1):
- El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez, Tlalpan, Mexico City, Mexico

REFERENCES:
- [Result] Nader-Kawachi J, Gongora-Rivera F, Santos-Zambrano J, Calzada P, Rios C. Neuroprotective effect of dapsone in patients with acute ischemic stroke: a pilot study. Neurol Res. 2007 Apr;29(3):331-4. doi: 10.1179/016164107X159234. PMID 17509235